CLINICAL TRIAL: NCT06297759
Title: The Validity and Reliability Study of Turkish Version of the Sense of Competence in Dementia Care Staff (SCIDS) Scale
Status: Not yet recruiting | Type: Observational
Sponsor: Yeditepe University (Other)
Collaborators: Acibadem University (Other)
Responsible Party: Sponsor
Other Study IDs: ATADEK-2023/16
Record Dates: First submitted 2024-03-01; First posted 2024-03-07 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Dementia
Keywords: dementia; Turkish version; dementia care staff; sense of competence in dementia care staff scale; validity; reliability
MeSH Terms: conditions — Dementia | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- healthcare professionals who care for patients with dementia: Participants will be selected by healthcare professionals who care for patients with dementia. At the first meeting, participants will be informed about the study, will be screened for inclusion criteria, and a written informed consent form will be obtained before testing.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Sense of Competence in Dementia Care Staff (SCIDS) Scale

SUMMARY:
The purpose of the study is to adapt the SCIDS into the Turkish version and validate it in the social and cultural context of Turkey to assess staff competency in dementia care in the long-term care setting.

DETAILED DESCRIPTION:
Most existing tools measuring care adequacy are targeted at family caregivers. Tools targeting formal dementia carers have focused primarily on dementia care knowledge, care attitudes and care workloads separately. There is less research investigating the assessment of competence in dementia care among formal healthcare staffs. There is no validated tool to accurately assess staff competency in dementia care in the long-term care setting in Turkey. Schepers et al. developed a scale dedicated to assessing Sense of Competence in Dementia Care Staff, including relationship building, maintaining personality, professionalism, and care challenges. Today, the scale has been used to evaluate the effectiveness of training programs and has demonstrated its applicability.

ELIGIBILITY:
Inclusion Criteria:

* Working as a dementia care staff for at least 1 year

Exclusion Criteria:

* Not volunteering

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Working as a dementia care staff in Acıbadem Health Group
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-06-10 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Sense of Competence in Dementia Care Staff Scale | Change from Baseline Scores at one week
  This scale includes competence in the field of dementia clinical practice, knowledge, skills and attitudes regarding dementia care.
  Scoring All items are scored from 1 (Not at all) to 4 (Very much). Higher scores mean a higher level of sense of confidence.
  Scores are added up for items from 1 to 17 for the overall SOCID-S score (ranging from 17 to 68) and for the subscales as follows:
  Professionalism: 7, 8, 9, 10, 12 (scores ranging from 5 to 20); Building Relationships: 1, 2, 3, 4 (scores ranging from 4 to 12); Care Challenges: 13, 14, 15, 17 (scores ranging from 4 to 12); and Sustaining Personhood: 5, 6, 11, 16 (scores ranging from 4 to 12)

SECONDARY OUTCOMES:
Caring Behaviors Inventory-24 | Change from Baseline Scores at one week
  Its correlation with Sense of Efficacy in Dementia Care Personnel will be conducted for construct validity.
  Assurance (8 items = 16, 17, 18, 20, 21, 22, 23, 24), knowledge-skill (5 items = 9, 10, 11, 12, 15), being respectful (6 items = 1, 3, It consists of 4 subgroups and 24 items: 5, 6, 13, 19) and commitment (5 items = 2, 4, 7, 8, 14), and a 6-point Likert-type scale (1 = never, 2 = almost never, 3=sometimes, 4=usually, 5=most of the time, 6=always) is used for the responses.
  As the subscale and total scale scores increase, the level of care quality perception of patients or nurses increases.

IPD SHARING:
Plan to Share IPD: Undecided